CLINICAL TRIAL: NCT00229411
Title: Experimental Like Observational Study of Teamwork Improvement in Multidisciplinary Intensive Care Team Before and After Simulation Training.
Brief Title: Simulation Training as a Tool for Teamwork Improvement in Multidisciplinary Intensive Care Team
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: SHEBA-05-3710-AN-CTIL
Record Dates: First submitted 2005-09-26; First posted 2005-09-29 (Estimated); Last update posted 2007-01-24 (Estimated); Status verified 2007-01

CONDITIONS: Education, Health
Keywords: intensive care; teamwork; medical errors; education; simulation
MeSH Terms: conditions — Health Education

INTERVENTIONS:
Behavioral: simulation training

SUMMARY:
The purpose of the study is to check whether training mixed teams of physicians and nurses from intensive care units on patient simulators improves teamwork within the teams.

DETAILED DESCRIPTION:
Patient safety and the prevention of medical error are primary goals of healthcare organizations. One of the means of reducing such errors is teamwork improvement. Simulation training, using advanced patient simulators, has been shown to improve diagnostic, resuscitation and technical skills amongst physicians and nurses. We intend to compare simulation training of a mixed team of physicians and nurses, using specifically designed scenarios based on real life experience, to frontal teaching sessions designed to enhance teamwork, by assessing teamwork, using accepted behavioral scales, during routine work, before and after both interventions.

ELIGIBILITY:
Inclusion Criteria:

* intensive care physicians and nurses working in respiratory ICU willing to participate in the study

Exclusion Criteria:

* unwilling to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2006-01; Study Completion 2006-05

PRIMARY OUTCOMES:
improvement in teamwork parameters as measured by previously published tools

CONTACTS AND LOCATIONS:
Overall Officials: Asaph E Nini, MD, Principal Investigator — Sheba Medical Center and Medical Simulation Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel